CLINICAL TRIAL: NCT05806021
Title: The Efficacy of Intra-articular Triamcinolone Acetonide 5mg vs. 10 mg vs. 40 mg in Patients With Knee Osteoarthritis: a Non-inferiority Randomized Controlled Double-blind Study
Brief Title: The Efficacy of Intra-articular Triamcinolone Acetonide 5mg vs. 10 mg vs. 40 mg in Patients With Knee Osteoarthritis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21.411
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Primary Gonarthrosis
Keywords: corticosteroid injection; minimal dose; non-inferiority
MeSH Terms: interventions — Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A TA 40 mg (Experimental): intra-articular injection of 40 mg of triamcinolone acetonide, which is the standard dose used
  Interventions: Drug: Triamcinolone Acetonide
- Group B TA 10 mg (Active Comparator): intra-articular injection of 10 mg of triamcinolone acetonide
  Interventions: Drug: Triamcinolone Acetonide
- Group C TA 5 mg (Active Comparator): intra-articular injection of 5 mg of triamcinolone acetonide
  Interventions: Drug: Triamcinolone Acetonide

INTERVENTIONS:
Drug: Triamcinolone Acetonide — Intra-articular injection. For each group, the total injected will be 3 ml. For syringes containing triamcinolone acetonide, the missing volume will be filled with 0.9% isotonic saline
  Other Names: Kenalog

SUMMARY:
Osteoarthritis of the knee is a common problem that is increasing in prevalence as the population ages. In a knee with osteoarthritis, there is variable damage to the articular cartilage and underlying bone that can cause varying degrees of pain. When pain is bothersome, osteoarthritis is treated to improve functional abilities.

One of the most recognized and used treatments is intra-articular cortisone injection. Cortisone is a powerful anti-inflammatory drug that is used to reduce pain.

Unfortunately, cortisone can have significant side effects, even when injected locally. The frequency and intensity of these side effects depend largely on the total dose injected. The main side effects include increased blood sugar levels, increased blood pressure and a temporary decrease in the secretion of the stress hormone, cortisol. In the long term, a decrease in articular cartilage thickness in the injected join and overall bone density reduction is also reported.

Despite many years of routine use, the smallest effective dose of cortisone injected into the knee joint is unknown.

The main objective of the study is to determine the impact on pain and function of different doses of cortisone injected into the knee. The cortisone chosen for this study is triamcinolone acetonide (TA).

DETAILED DESCRIPTION:
Gonarthrosis is a very prevalent condition affecting especially people over the age of 60 years old. It is a major cause of pain and functional impairment in Canada. The prevalence and associated economic burden continue to increase.

Despite the prevalence of this condition, the management of symptomatic gonarthrosis remains a controversial subject. Multiple treatment alternatives are available, none of which has been proven to be superior to the others beyond any doubt. However, certain therapeutic modalities are better recognized and more frequently used, such as intra-articular corticosteroid injections. In 2022, an expert consensus review of the available literature concluded that the use of intra-articular corticosteroids is effective in the treatment of symptomatic gonarthrosis. This is also the conclusion of the most recent American College of Rheumatology (ACR) guideline, which "strongly recommends" the use of this type of injection in gonarthrosis .

Despite decades of use, there is insufficient evidence to recommend a specific type and dose of corticosteroid. The choice of cortisone type in the usual practice of physicians performing intra-articular knee infiltrations is therefore based on experience and the biochemical properties of the different cortisones. Those with larger particles due to esterification of the corticoid, such as triamcinolone acetonide (TA) and methylprednisolone acetate, are known to have a longer duration of action. They are therefore the two most frequently used in studies on the subject. The dose used is based on historical use and is not, to our knowledge, based on any fundamental evidence. This dose of TA injected into a joint is usually 40 mg. Some authors have shown us that it is not useful to inject higher doses than this into a knee because increasing the dose does not improve the outcome of the injection. However, there was no literature related to the minimally effective intra-articular TA dose in the knee, until recently. Indeed, Utamawatin et al. recently reported that 10mg of TA did not appear to be less effective than 40mg when injected into knees with primary osteoarthritis.

This minimally effective dose is important because side effects associated with cortisone use have been reported. The adverse effects of oral corticosteroids are better known and documented than intra-articular ones. By a mechanism that is only partially elucidated, intra-articular infiltrations can produce the same systemic effects as oral. Habib et al. reports that systemic side effects increase with the concentration and time of exposure to the substance. To our knowledge, the minimal dose of intra-articular corticosteroid to produce a systemic effect is not documented.

Systemic effects occur in multiple systems. They affect several metabolisms such as glucose, gastrointestinal, lipid, adipose tissue, bone, immune, cardiovascular, sex hormones and the hypothalamic-pituitary axis. The mood can also be affected.

Thus, intra-articular infiltrations can cause both local and systemic problems that are directly related to the dose injected.

PRIMARY OBJECTIVE

○ To demonstrate the non-inferiority of a 10 mg and 5 mg intra-articular corticosteroid injection compared to the standard 40 mg dose on patient function at 1 month post-injection.

SECONDARY OBJECTIVES

* To demonstrate the non-inferiority of a 10 mg and 5 mg intra-articular corticosteroid injection compared to the standard 40 mg dose on patient function at 2, 3 and 6 months post-injection.
* To demonstrate the non-inferiority of a 10 mg and 5 mg intra-articular corticosteroid injection compared to the standard 40 mg dose on pain and stiffness in patients at 1, 2, 3 and 6 months post-injection.
* To know the patient's satisfaction with the treatment at 3 and 6 month post-injection METHODOLOGY Type of study

  * Randomized clinical trial
  * Non-inferiority study Recruiting
  * Outpatient clinic of the physiatry, rheumatology or orthopedics departments of the University of Montreal Hospital.

Participants

* Patients referred to physiatry for symptomatic primary gonarthrosis
* Physiatrists will complete a history and physical examination for each participant.

Randomization of participants

* Patients meeting the study inclusion criteria will be randomized into one of the three groups
* Group allocation will be done randomly by computer. The mechanism for running the allocation sequence for randomization will be with RedCAP software.
* Physiatrists evaluating outcomes, participants, and data analysis will be blinded.
* Syringes will be preassembled by someone external to the study. The syringes will be covered with opaque paper. The contents of the latter will therefore not be visible to the participant or the physician performing the procedure.
* Participants will be able to know at the end of the study in which group they were allocated.

Intervention

* For ethical reasons, considering the superiority of cortisone injections in the latest international recommendations, it was decided not to use a placebo group.
* All eligible patients will have a standing radiograph with weight-bearing anteroposterior view, lateral view, and patellar view that will be done at CHUM, unless a recent radiograph done at another center is available for review by a CHUM radiologist. This is to obtain standardized imaging results for our study.
* The technique of the procedure is done according to the practical guide Malanga and Mautner: Atlas of Ultrasound-Guided Musculoskeletal Injections.
* Ultrasound guidance will be used for all intra-articular knee injections. Canon I-700 ultrasound machine.
* Patients will be placed in the supine position with the knee resting on a towel for slight flexion.
* The procedure is performed under sterile conditions.
* The skin is disinfected with a CHUM-approved chlorhexidine-based product.
* The ultrasound probe is disinfected with an approved disinfectant product.
* With a sterile gel on the skin, the probe is positioned short-axis over the distal quadricipital tendon.
* The supra-patellar recess is visualized between the prefemoral fat pad posteriorly and the suprapatellar fat pad anteriorly as an area containing hypoechoic or anechoic fluid.
* If there is a significant intra-articular effusion, the fluid will by removed via punture prior to injection. This information will be noted on a sheet including the total volume removed.
* On the lateral border of the knee with an approach parallel to the probe, a 3ml syringe mounted on a 25G needle (or 18-20G if prior puncture) is inserted. A dermal point with 1% xylocaine will be made before the injection if prior puncture given the use of a larger needle gauge.
* In real time under ultrasound guidance, the needle is advanced from lateral to medial towards the supra-patellar recess.
* Once the needle is properly positioned in the recessus, the physiatrist injects the contents of the pre-mounted 3ml syringe.
* If there is no visible fluid in the supra-patellar recess, the medial mid-patellar region is targeted. This technique is not influenced by the presence or absence of effusion. The probe is placed in a short axis on the knee with the patella superior and the medial femoral condyle inferior. The joint space is located between the two structures under the patellar retinaculum. The needle is advanced parallel to the probe from medial to lateral to penetrate the joint space. This technique can also be performed lateral to the knee at the discretion of the physiatrist.
* After the injection, it is recommended to apply a cold water compress or ice to the injection site 5-10 min which can be repeated 3 to 4 times during the day in case of pain. Acetaminophen may be taken to reduce discomfort following the injection.
* All techniques under ultrasound guidance will be performed by a physiatrist trained in musculoskeletal ultrasound.
* Intra-articular cortisone infiltration is not the only treatment for gonarthrosis. Therefore, all patients will have as a recommendation some of the non-pharmacologic recommendations mentioned in the ACR8 guide.
* Patients will be suggested not to add other treatment modalities to avoid biasing the results such as orthotic, acupuncture, massage, anti-inflammatory or other medications, other injectable treatments etc. If the patient is already wearing an orthosis, he/she can continue to wear it.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic primary gonarthrosis of over 6 months duration (gonarthrosis according to the American College of Rheumatology criteria)
* Grade 1 to 3 Kellgren-Lawrence femorotibial osteoarthritis
* Knee pain provoked by activity over 4 and under 8 on 10 (Visual Analog Scale)

Exclusion Criteria:

* Bilateral symptomatic primary gonarthrosis
* Grade 4 Kellgren-Lawrence femorotibial osteoarthritis
* Isolated patellofemoral osteoarthritis
* Intra-articular corticosteroid infiltration to the knee within the past 3 months or chronic use of per os corticosteroid
* Intra-articular hyaluronic acid infiltration within the past 12 months.
* Intra-articular infiltration of platelet-rich plasma within the past 12 months.
* Disease affecting the study joint (systemic inflammatory disease, history of septic arthritis, osteonecrosis, etc.).
* Suspicion or presence of active local infectious process.
* Presence or suspicion of local neoplasia or metastasis
* Recent severe trauma to the knee (≤ 3 months)
* Significant cognitive impairment or inadequate language proficiency not allowing adequate response to study questionnaires
* Any other serious medical condition that does not allow participation in the study or may be a contraindication to cortisone injection

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 327 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
WOMAC Function | 1 month post-injection
  Western Ontario and McMaster Universities Osteoarthritis index (WOMAC), FUNCTION sub-score.
  The WOMAC is a 24-item questionnaire subdivided into three sections. It includes 5 items related to pain, 2 items related to stiffness, and 17 items related to physical function. Only function section will be used as the primary outcome measure. Responses to each of the 17 questions will be scored on graduated scales from 0 to 10 where 0 means no pain and 10 means the worst possible pain. Higher scores indicate greater symptom intensity. A total score out of a maximum of 68 points for function will be compiled and used for statistical analysis.

SECONDARY OUTCOMES:
WOMAC Total | 1, 2, 3 and 6 months post-injection
  Western Ontario and McMaster Universities Osteoarthritis index (WOMAC), TOTAL score.
  The WOMAC is a 24-item questionnaire subdivided into three sections. It includes 5 items related to pain, 2 items related to stiffness, and 17 items related to physical function. All three item sections (pain, function, stiffness) will be used. Responses to each of the 24 questions will be scored on graduated scales from 0 to 10 where 0 means no pain and 10 means the worst possible pain. Higher scores indicate greater symptom intensity. A total score out of a maximum of 96 points as well as sectional scores (pain out of 20, function out of 68 and stiffness out of 8) will be compiled and used for statistical analysis. The WOMAC provides reliable scores that are highly sensitive to changes in pain and function in people with osteoarthritis.
VAS | 1, 2, 3 and 6 months post-injection
  Visual analog pain scale (1-10). The visual analogue scale consists of a graduated scale from 0 to 10 where 0 means no pain and 10 means the worst possible pain. This scale will be used to document the intensity of the pain
LIKERT | 3 and 6 months post-injection
  Likert subjective satisfaction scale (1-5)

CONTACTS AND LOCATIONS:
Overall Officials: Dien Hung Luong, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier Universitaire de Montréal - Hôtel-Dieu, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sharma L. Osteoarthritis of the Knee. N Engl J Med. 2021 Jan 7;384(1):51-59. doi: 10.1056/NEJMcp1903768. No abstract available. PMID 33406330
- [Background] Khan M, Bhandari M. Cochrane in CORR(R): Intra-articular Corticosteroid For Knee Osteoarthritis. Clin Orthop Relat Res. 2018 Jul;476(7):1391-1392. doi: 10.1097/CORR.0000000000000358. No abstract available. PMID 29846205
- [Background] Hunter CW, Deer TR, Jones MR, Chang Chien GC, D'Souza RS, Davis T, Eldon ER, Esposito MF, Goree JH, Hewan-Lowe L, Maloney JA, Mazzola AJ, Michels JS, Layno-Moses A, Patel S, Tari J, Weisbein JS, Goulding KA, Chhabra A, Hassebrock J, Wie C, Beall D, Sayed D, Strand N. Consensus Guidelines on Interventional Therapies for Knee Pain (STEP Guidelines) from the American Society of Pain and Neuroscience. J Pain Res. 2022 Sep 8;15:2683-2745. doi: 10.2147/JPR.S370469. eCollection 2022. PMID 36132996
- [Background] HOLLANDER JL. Intra-articular hydrocortisone in arthritis and allied conditions; a summary of two years' clinical experience. J Bone Joint Surg Am. 1953 Oct;35-A(4):983-90. No abstract available. PMID 13108900
- [Background] HOLLANDER JL, BROWN EM Jr, JESSAR RA, BROWN CY. Hydrocortisone and cortisone injected into arthritic joints; comparative effects of and use of hydrocortisone as a local antiarthritic agent. J Am Med Assoc. 1951 Dec 22;147(17):1629-35. doi: 10.1001/jama.1951.03670340019005. No abstract available. PMID 14880415
- [Background] Johnston PC, Lansang MC, Chatterjee S, Kennedy L. Intra-articular glucocorticoid injections and their effect on hypothalamic-pituitary-adrenal (HPA)-axis function. Endocrine. 2015 Mar;48(2):410-6. doi: 10.1007/s12020-014-0409-5. Epub 2014 Sep 3. PMID 25182149
- [Background] Kolasinski SL, Neogi T, Hochberg MC, Oatis C, Guyatt G, Block J, Callahan L, Copenhaver C, Dodge C, Felson D, Gellar K, Harvey WF, Hawker G, Herzig E, Kwoh CK, Nelson AE, Samuels J, Scanzello C, White D, Wise B, Altman RD, DiRenzo D, Fontanarosa J, Giradi G, Ishimori M, Misra D, Shah AA, Shmagel AK, Thoma LM, Turgunbaev M, Turner AS, Reston J. 2019 American College of Rheumatology/Arthritis Foundation Guideline for the Management of Osteoarthritis of the Hand, Hip, and Knee. Arthritis Care Res (Hoboken). 2020 Feb;72(2):149-162. doi: 10.1002/acr.24131. Epub 2020 Jan 6. PMID 31908149
- [Background] Shah A, Mak D, Davies AM, James SL, Botchu R. Musculoskeletal Corticosteroid Administration: Current Concepts. Can Assoc Radiol J. 2019 Feb;70(1):29-36. doi: 10.1016/j.carj.2018.11.002. PMID 30691559
- [Background] Cushman DM, Bruno B, Christiansen J, Schultz A, McCormick ZL. Efficacy of Injected Corticosteroid Type, Dose, and Volume for Pain in Large Joints: A Narrative Review. PM R. 2018 Jul;10(7):748-757. doi: 10.1016/j.pmrj.2018.01.002. Epub 2018 Jan 31. PMID 29407227
- [Background] Cushman DM, Ofek E, Syed RH, Clements N, Gardner JE, Sams JM, Mulvey JL, McCormick ZL. Comparison of Varying Corticosteroid Type, Dose, and Volume for the Treatment of Pain in Small- and Intermediate-Size Joint Injections: A Narrative Review. PM R. 2019 Jul;11(7):758-770. doi: 10.1016/j.pmrj.2018.09.040. Epub 2019 Jun 5. PMID 31166662
- [Background] Utamawatin K, Phruetthiphat OA, Apinyankul R, Chaiamnuay S. The efficacy of intra-articular triamcinolone acetonide 10 mg vs. 40 mg in patients with knee osteoarthritis: a non-inferiority, randomized, controlled, double-blind, multicenter study. BMC Musculoskelet Disord. 2023 Feb 3;24(1):92. doi: 10.1186/s12891-023-06191-6. PMID 36737698
- [Background] Kim KH, Park JW, Kim SJ. High- vs Low-Dose Corticosteroid Injection in the Treatment of Adhesive Capsulitis with Severe Pain: A Randomized Controlled Double-Blind Study. Pain Med. 2018 Apr 1;19(4):735-741. doi: 10.1093/pm/pnx227. PMID 29117299
- [Background] Stout A, Friedly J, Standaert CJ. Systemic Absorption and Side Effects of Locally Injected Glucocorticoids. PM R. 2019 Apr;11(4):409-419. doi: 10.1002/pmrj.12042. Epub 2019 Mar 29. PMID 30925034
- [Background] Habib GS. Systemic effects of intra-articular corticosteroids. Clin Rheumatol. 2009 Jul;28(7):749-56. doi: 10.1007/s10067-009-1135-x. Epub 2009 Feb 28. PMID 19252817
- [Background] Habib GS, Bashir M, Jabbour A. Increased blood glucose levels following intra-articular injection of methylprednisolone acetate in patients with controlled diabetes and symptomatic osteoarthritis of the knee. Ann Rheum Dis. 2008 Dec;67(12):1790-1. doi: 10.1136/ard.2008.089722. No abstract available. PMID 19005159
- [Background] Choudhry MN, Malik RA, Charalambous CP. Blood Glucose Levels Following Intra-Articular Steroid Injections in Patients with Diabetes: A Systematic Review. JBJS Rev. 2016 Mar 22;4(3):e5. doi: 10.2106/JBJS.RVW.O.00029. PMID 27500431
- [Background] Habib GS, Miari W. The effect of intra-articular triamcinolone preparations on blood glucose levels in diabetic patients: a controlled study. J Clin Rheumatol. 2011 Sep;17(6):302-5. doi: 10.1097/RHU.0b013e31822acd7c. PMID 21869712
- [Background] Taliaferro K, Crawford A, Jabara J, Lynch J, Jung E, Zvirbulis R, Banka T. Intraocular Pressure Increases After Intraarticular Knee Injection With Triamcinolone but Not Hyaluronic Acid. Clin Orthop Relat Res. 2018 Jul;476(7):1420-1425. doi: 10.1007/s11999.0000000000000261. PMID 29533245
- [Background] Wernecke C, Braun HJ, Dragoo JL. The Effect of Intra-articular Corticosteroids on Articular Cartilage: A Systematic Review. Orthop J Sports Med. 2015 Apr 27;3(5):2325967115581163. doi: 10.1177/2325967115581163. eCollection 2015 May. PMID 26674652
- [Background] McAlindon TE, LaValley MP, Harvey WF, Price LL, Driban JB, Zhang M, Ward RJ. Effect of Intra-articular Triamcinolone vs Saline on Knee Cartilage Volume and Pain in Patients With Knee Osteoarthritis: A Randomized Clinical Trial. JAMA. 2017 May 16;317(19):1967-1975. doi: 10.1001/jama.2017.5283. PMID 28510679
- [Background] Wheeler SG. Steroid Knee Injections for Arthritis Are No Better than Placebo in a Randomized Controlled Trial. J Gen Intern Med. 2020 Oct;35(10):3137-3139. doi: 10.1007/s11606-020-05647-y. No abstract available. PMID 32556876
- [Background] Schneider BJ, Mattie R, Smith C. Cumulative Lifetime Steroid Exposure via Epidural Administration. Pain Med. 2019 Nov 1;20(11):2323-2324. doi: 10.1093/pm/pnz203. No abstract available. PMID 31504872
- [Background] Altman R, Asch E, Bloch D, Bole G, Borenstein D, Brandt K, Christy W, Cooke TD, Greenwald R, Hochberg M, et al. Development of criteria for the classification and reporting of osteoarthritis. Classification of osteoarthritis of the knee. Diagnostic and Therapeutic Criteria Committee of the American Rheumatism Association. Arthritis Rheum. 1986 Aug;29(8):1039-49. doi: 10.1002/art.1780290816. PMID 3741515
- [Background] Kohn MD, Sassoon AA, Fernando ND. Classifications in Brief: Kellgren-Lawrence Classification of Osteoarthritis. Clin Orthop Relat Res. 2016 Aug;474(8):1886-93. doi: 10.1007/s11999-016-4732-4. Epub 2016 Feb 12. No abstract available. PMID 26872913
- [Background] Dworkin RH, Turk DC, Farrar JT, Haythornthwaite JA, Jensen MP, Katz NP, Kerns RD, Stucki G, Allen RR, Bellamy N, Carr DB, Chandler J, Cowan P, Dionne R, Galer BS, Hertz S, Jadad AR, Kramer LD, Manning DC, Martin S, McCormick CG, McDermott MP, McGrath P, Quessy S, Rappaport BA, Robbins W, Robinson JP, Rothman M, Royal MA, Simon L, Stauffer JW, Stein W, Tollett J, Wernicke J, Witter J; IMMPACT. Core outcome measures for chronic pain clinical trials: IMMPACT recommendations. Pain. 2005 Jan;113(1-2):9-19. doi: 10.1016/j.pain.2004.09.012. No abstract available. PMID 15621359
- [Background] Sullivan GM, Artino AR Jr. Analyzing and interpreting data from likert-type scales. J Grad Med Educ. 2013 Dec;5(4):541-2. doi: 10.4300/JGME-5-4-18. No abstract available. PMID 24454995
- [Background] Tarhan S, Unlu Z. Magnetic resonance imaging and ultrasonographic evaluation of the patients with knee osteoarthritis: a comparative study. Clin Rheumatol. 2003 Sep;22(3):181-8. doi: 10.1007/s10067-002-0694-x. PMID 14505208
- [Background] Messier SP, Resnik AE, Beavers DP, Mihalko SL, Miller GD, Nicklas BJ, deVita P, Hunter DJ, Lyles MF, Eckstein F, Guermazi A, Loeser RF. Intentional Weight Loss in Overweight and Obese Patients With Knee Osteoarthritis: Is More Better? Arthritis Care Res (Hoboken). 2018 Nov;70(11):1569-1575. doi: 10.1002/acr.23608. PMID 29911741
- [Background] Salaffi F, Stancati A, Silvestri CA, Ciapetti A, Grassi W. Minimal clinically important changes in chronic musculoskeletal pain intensity measured on a numerical rating scale. Eur J Pain. 2004 Aug;8(4):283-91. doi: 10.1016/j.ejpain.2003.09.004. PMID 15207508
- [Background] Bellamy N, Hochberg M, Tubach F, Martin-Mola E, Awada H, Bombardier C, Hajjaj-Hassouni N, Logeart I, Matucci-Cerinic M, van de Laar M, van der Heijde D, Dougados M. Development of multinational definitions of minimal clinically important improvement and patient acceptable symptomatic state in osteoarthritis. Arthritis Care Res (Hoboken). 2015 Jul;67(7):972-80. doi: 10.1002/acr.22538. PMID 25581339
- [Background] Seror P, Pluvinage P, d'Andre FL, Benamou P, Attuil G. Frequency of sepsis after local corticosteroid injection (an inquiry on 1160000 injections in rheumatological private practice in France). Rheumatology (Oxford). 1999 Dec;38(12):1272-4. doi: 10.1093/rheumatology/38.12.1272. PMID 10587558
- [Background] Manchikanti L, Cash KA, Pampati V, Damron KS, McManus CD. Evaluation of lumbar transforaminal epidural injections with needle placement and contrast flow patterns: a prospective, descriptive report. Pain Physician. 2004 Apr;7(2):217-23. PMID 16868595
- [Background] Friedman DM, Moore ME. The efficacy of intraarticular steroids in osteoarthritis: a double-blind study. J Rheumatol. 1980 Nov-Dec;7(6):850-6. PMID 7009857
- [Background] Pattrick M, Doherty M. Facial flushing after intra-articular injection of steroid. Br Med J (Clin Res Ed). 1987 Nov 28;295(6610):1380. doi: 10.1136/bmj.295.6610.1380. No abstract available. PMID 3121023
- [Background] Gitkind AI, Shah B, Thomas M. Epidural corticosteroid injections as a possible cause of menorrhagia: a case report. Pain Med. 2010 May;11(5):713-5. doi: 10.1111/j.1526-4637.2009.00775.x. Epub 2010 Jan 8. PMID 20070546
- [Background] Suh-Burgmann E, Hung YY, Mura J. Abnormal vaginal bleeding after epidural steroid injection: a paired observation cohort study. Am J Obstet Gynecol. 2013 Sep;209(3):206.e1-6. doi: 10.1016/j.ajog.2013.06.045. Epub 2013 Jun 28. PMID 23816843
- See also: Outcome scale description — https://www.orthobullets.com/basic-science/9087/outcome-measure-tool